CLINICAL TRIAL: NCT01619046
Title: Determination of Safety, Efficacy and Pharmacokinetics of GreenGene™ F in Previously Treated Patients 12 Years of Age or Older Diagnosed With Severe Hemophilia A
Brief Title: Safety, Efficacy and Pharmacokinetics of GreenGene™ F to Previously Treated Patients With Severe Hemophilia A
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Green Cross Corporation (Industry)
Collaborators: Atlantic Research Group (Other)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GreenGeneF_P3
Record Dates: First submitted 2012-05-31; First posted 2012-06-14 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-07

CONDITIONS: Hemophilia A
Keywords: GreenGene™F, Previously Treated Patients
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- PK substudy (Active Comparator): A cohort of 13-18 subjects will be included in the pharmacokinetic (PK) evaluation of GreenGene™ F and an approved recombinant Factor VIII product (Refacto AF); a minimum of 13 of these subjects will be re-evaluated at study end (50 exposure day).
  Interventions: Biological: GreenGene™ F and an approved recombinant Factor VIII product
- Prophylaxis safety and efficacy substudy (Experimental): Hemostatic efficacy of GreenGene™ F will be assessed by its effectiveness in controlling spontaneous or traumatic bleeding episodes and by the rate of breakthrough bleeding during prophylaxis over ≥ 50 exposure days.
  Interventions: Biological: GreenGene™ F
- On-demand safety and efficacy substudy (Experimental): Hemostatic efficacy of GreenGene™ F will be assessed by its effectiveness in controlling spontaneous or traumatic bleeding episodes and by the rate of breakthrough bleeding in a minimum of 10 on demand treated subjects during 50 exposure days.
  Interventions: Biological: GreenGene™ F
- Surgical substudy (Experimental): Peri-operative hemostatic control of GreenGene™ F in surgery or invasive procedures will be assessed in at least 10 surgeries, some of them major, in at least five subjects
  Interventions: Biological: GreenGene™ F

INTERVENTIONS:
Biological: GreenGene™ F and an approved recombinant Factor VIII product — one 50 IU/kg, intra-venous infusion over 5 minutes, Infusion rate < 10 mL/min
  Other Names: GreenGeneF; GreenGene F
  Arms: PK substudy
Biological: GreenGene™ F — intra-venous infusion, 30 ± 5 IU/kg infusions 3 times per week with dose escalation to 45 ± 5 IU/kg if appropriate, for 50 exposure days
  Other Names: GreenGeneF; GreenGene F
  Arms: Prophylaxis safety and efficacy substudy
Biological: GreenGene™ F — intra-venous infusion,
  On-demand safety and efficacy substudy:
  minor bleed = 10-20 IU/kg moderate bleed = 15-30 IU/kg major bleed = 30-50 IU/kg
  Other Names: GreenGeneF; GreenGene F
  Arms: On-demand safety and efficacy substudy
Biological: GreenGene™ F — intra venous infusion,
  Surgical substudy:
  Minor surgery including tooth extraction = Post in fusion FVIII level of 60-100% of normal. A single bolus infusion (30-50 IU/kg) beginning within one hour of the operation. Optional additional dosing every 12 to 24 hours as needed to control bleeding.
  Major surgery = Pre- and post infusion FVIII level 80-120% of normal. Preoperative bolus infusion: 40-60 IU/kg. Verified 100% activity prior to surgery. Maintenance bolus infusion (40-60 IU/kg) repeat infusions every 8 to 24 hours, depending on the desired level.
  Other Names: GreenGeneF; GreenGene F
  Arms: Surgical substudy

SUMMARY:
The purpose of this study is to assess the safety, efficacy and pharmacokinetics of GreenGene™ F in subjects with severe hemophilia A previously treated (> 150 exposure days) with a Factor VIII concentrate and without presence or history of inhibitors to FVIII (Factor VIII).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects age ≥ 12 years at the time of informed consent
2. Body weight ≥ 35 kg
3. Diagnosed with severe hemophilia A. All subjects must have severe hemophilia A with baseline FVIII <1% activity; <0.01 IU/mL
4. Have ≥ 150 previous exposure days to FVIII concentrates, as documented in the subject's medical records
5. Subjects included in the on-demand treatment cohort must have a verifiable record of at least three bleeding episodes per month on average in the last 6 months prior to enrollment
6. Negative assays for FVIII inhibitor at inclusion (<0.6BU Nijmegen assay)
7. Negative assays for FVIII inhibitor in subject files (<0.6BU Nijmegen assay) No history of positive inhibitor is allowed
8. Normal liver and kidney function.
9. Platelet count ≥ 100,000 μL
10. Normal prothrombin time or International Normalized Ratio (INR) < 1.5
11. Subjects receiving therapy for human immunodeficiency virus (HIV) or hepatitis must be on a stable treatment regimen
12. Subjects must be able to withhold FVIII infusions for approximately 72 h prior to each FVIII activity and inhibitor assay (96 h if participating in the PK sub study)
13. Absolute CD4 lymphocyte cell count ≥ 200 μL
14. Signed the written informed consent form or informed consent was obtained from the subject's legal guardian
15. Females must not be lactating or pregnant at Screening or Baseline (as documented by a negative beta-human chorionic gonadotropin [ß hCG] test with a minimum sensitivity of 25 IU/L or equivalent units of ß hCG). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug
16. All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group and without other known or suspected cause) or have been sterilized surgically (i.e. bilateral tubal ligation, total hysterectomy or bilateral oophorectomy, all with surgery at least one month before dosing)
17. Willing and able to comply with all aspects of the protocol

Exclusion Criteria:

1. Presence at Screening of FVIII inhibitor ≥ 0.6 BU as tested with the Nijmegen modification of the Bethesda assay in either central or local laboratory
2. History of FVIII inhibitor of ≥ 0.6 BU as measured using the Nijmegen modification of the Bethesda assay
3. History of FVIII inhibitor ≥ 1.0 BU if the subject has been tested routinely using the original Bethesda assay, or history of periods with low recovery and no response to Factor VIII treatment
4. Demonstrated an inability to respond to conventional doses of FVIII therapy
5. History of incremental recovery of Factor VIII <1.35% per IU/kg infused
6. Hematological disorders or blood coagulation diseases (e.g., idiopathic thrombocytopenic purpura, von Willebrand disease, etc.) other than hemophilia A
7. Laboratory or clinical evidence of portal vein hypertension including,(but not limited to, an INR > 1.4, the presence of splenomegaly and/or spider angiomata on physical examination and/or a history of esophageal hemorrhage or documented esophageal varices
8. Uncontrolled hypertension (diastolic blood pressure >100 mm Hg)
9. Hemoglobin < 10 g.dL
10. HIV disease symptoms regardless of presence of HIV antibodies
11. Routine administration (or planned routine administration during the course of the study), of immunosuppressive or immunomodulating drugs other than antiretroviral therapy (e.g., steroids, beta-interferon)
12. Severe renal dysfunction (creatinine > 2x upper limit of normal [ULN], total bilirubin > 2x the ULN)
13. Liver disease (alanine aminotransferase [ALT], aspartate aminotransferase [ AST] > 3x the ULN)
14. History of diabetes or other metabolic disease
15. History of hypersensitivity or serious adverse reaction to recombinant or plasma-derived FVIII concentrate
16. History of pretreatment prior to the administration of FVIII products (e.g., of antihistamines)
17. Regular use of antifibrinolytics or medications affecting platelet function
18. Hypersensitivity to hamster-or mouse derived proteins
19. Blood transfusions within 30 days of enrollment into the study
20. Current participation in another investigational drug or device study, or participated in a clinical study involving an investigational drug or device within 30 days of enrollment into the study
21. Unable or unwilling to cooperate with study procedures

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-07 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Number of subject with development of inhibitors | evert 3 months, up to 18 months
  Development of neutralizing antibodies (inhibitors) will be followed during the regular visits, average of 3 months.

SECONDARY OUTCOMES:
Describe the PK profile of GreenGene™ F | Pre-dose, 0~48hours post-dose
  AUC, AUMC, Half-life, Incremental recovery, Mean residence time (MRT), Clearance, Volume of distribution - steady state, Cmax, Tmax

CONTACTS AND LOCATIONS:
Overall Officials: Paul LeoFrancis Giangrande, MD, Principal Investigator — Oxford Haemophilic Centre and Thrombosis Unit, Churchill Hospital
Locations (34):
- United States (10):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Los Angeles Orthopaedic Hospital - Hemophilia Treatment Center, Los Angeles, California
  - Harbor - UCLA Pediatrics, Torrance, California
  - University of Miami - Comprehensive Hemophilia Center, Miami, Florida
  - St. Luke's Boise Medical Center, Boise, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Michigan State University Center for Bleeding Disorders & Clotting Disorders, East Lansing, Michigan
  - Children's Mercy Hospital - Kansas City Regional Hemophilia Center, Kansas City, Missouri
  - Long Island Jewish Medical Center - Hemophilia Treatment Center, New Hyde Park, New York
  - Oregon Health and Science University, Portland, Oregon
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - McMaster Children's Hospital, Hamilton, Ontario
- Research Associates, Ltd., Christchurch, New Zealand, New Zealand
- Poland (2):
  - Instytut Hematologii i Transfuzjologii, Warsaw
  - wojewodzki szpital Specjalistyczny, klinika hematologii uniwersytetu medycznego w łodzi, Łodzi
- Russia (5):
  - Barnaul Altai State Scientfic Center, Barnaul
  - Kirov Research Institute of Hematology and Blood Transfusion, Kirov
  - Ismailov City Children's Clinical Hospital of Board of Health of Moscow City, Moscow
  - State Budget Educational Institution of Higher professional Education "Samara State Medical University" of the Ministry of Health and Social Process of the Russian Federation, Samara
  - Ufa Republican Clinical Hospital, Ufa
- Ukraine (6):
  - Dnepropetrovsk City Clinical Hospital, Dnipro
  - Institute of Urgent and Reconstructive surgery named after V.K. Gusak of National Academy of Medical Sciences of Ukraine, Donetsk
  - Kharkov Regional Clinical Oncology Center, Kharkiv
  - Kyiv City Clinical Hospital No 91, Kyiv
  - Institute of Blood Pathology and Transfusion Medicine of National Academy of Medical Sciences of Ukraine Department of Surgery and Clinical Transfusiology, Lviv
  - Zaporizhzhya Region Clinical Child Hospital, Zaporzhye
- United Kingdom (8):
  - Royal Cornwall Hospital, Department of Haematology, Truro, Cornwall
  - Hull Haemophillia Centre, Hull Royal Infirmary, Humberside, Hull
  - Central Manchester University Hospitals, Manchester, Lancashire
  - St. Thomas' Hospital, City of Westminster, London
  - North Hampshire Haemophilia Centre, Basingstoke, North Hampshire
  - University of Liverpool, Liverpool
  - Royal Free Hospital, Haemophilia Centre & Thrombosis Unit, London
  - Churchill Hospital, Oxford, Oxford